CLINICAL TRIAL: NCT02609464
Title: The Use of Barbed Sutures in Total Hip Arthroplasty: A Prospective, Randomized, and Controlled Clinical Trial
Brief Title: The Use of Barbed Sutures in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15P01
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Inturrupted Knotte Sutures (Active Comparator)
  Interventions: Device: Interrupted Knotted Sutures
- Barbed Sutures (Active Comparator)
  Interventions: Device: STRATAFIX Symmetric PDS PLUS Knotless Tissue Control Devices

INTERVENTIONS:
Device: Interrupted Knotted Sutures
  Arms: Inturrupted Knotte Sutures
Device: STRATAFIX Symmetric PDS PLUS Knotless Tissue Control Devices
  Arms: Barbed Sutures

SUMMARY:
The purpose of this study is to evaluate the role of new barbed suture for closure of wound during total hip arthroplasty in reducing the risk for wound healing problems.

ELIGIBILITY:
Inclusion criteria:

* All patients receiving elective primary THA through the direct anterior approach, treated by the primary investigator (JP) at the Thomas Jefferson University Hospital or Rothman Specialty Hospital.

Exclusion Criteria:

* Prior surgical incision or scar in close proximity of the proposed incision (<2 cm).
* Local skin conditions such as dermatitis, eczema, or psoriasis.
* Active or previous infection in the skin or the hip.
* Inflammatory arthritis; connective tissue or vascular disorders or diseases that would adversely affect wound healing including the use of oral or topical cortico-steroid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of suture abscess or other wound related compilation | Within 30 days of surgery